CLINICAL TRIAL: NCT00023764
Title: Phase II Study of PS-341 in Low Grade Lymphoproliferative Disorders
Brief Title: Bortezomib in Treating Patients With Lymphoproliferative Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01406; NCI-2012-01406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UNMC-03903; MSKCC-01049; NCI-2795; CDR0000068860; CWRU-MSKCC-1Y02; 01-049 (Other: Memorial Sloan-Kettering Cancer Center); 2795 (Other: CTEP); P30CA008748 (NIH); U01CA062502 (NIH); N01CM62206 (NIH)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Results first posted 2014-04-01 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Bortezomib

ARMS (1):
- Arm I (Experimental): Patients receive an infusion of bortezomib (dose of 1.8 mg/m2) over 3-5 seconds once weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve at least a partial response lasting at least 6 months may receive retreatment.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
Phase II trial to study the effectiveness of bortezomib in treating patients who have low-grade lymphoproliferative disorders. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the frequency and duration of complete and partial response rates in patients with grade I, II, or III follicular lymphoma or mantle cell lymphoma treated with bortezomib.

SECONDARY OBJECTIVES:

I. Determine the response of minimal residual disease by polymerase chain reaction (PCR) detectable or clonotypic PCR minimal residual disease in bone marrow of patients treated with this regimen.

II. Determine the time to progression and overall survival of patients treated with this regimen.

III. Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients are stratified according to disease type (follicular lymphoma vs mantle cell lymphoma).

Patients receive an infusion of bortezomib over 3-5 seconds once weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve at least a partial response lasting at least 6 months may receive retreatment.

Patients are followed every 3 months for 1 year and then every 4 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed lymphoproliferative disorder of 1 of the following subtypes:
* * Relapsed or refractory grade I, II, or III follicular center cell lymphoma

  * Relapsed or refractory mantle cell lymphoma
* Measurable disease for non-Hodgkin's lymphoma (NHL) only

  * At least 1 unidimensionally measurable lesion
  * At least 2 cm by conventional techniques OR at least 1 cm by spiral CT scan
  * Lymph nodes no greater than 1 cm in short axis considered normal
* Absolute lymphocytosis greater than 5,000/mm^3 with B-cell phenotype (CD19, 20,or 23 positive) with more than 30% bone marrow lymphocytes for CLL or other leukemic forms of NHL
* No known brain metastases
* Performance status - Karnofsky 70-100%
* At least 3 months
* See Disease Characteristics
* Absolute neutrophil count greater than 1,500/mm^3 (500/mm^3 if lymphomatous involvement of bone marrow)
* Platelet count greater than 50,000/mm^3
* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN (4 times ULN in case of liver metastases)
* Creatinine less than 1.5 times ULN
* No symptomatic congestive heart failure
* No New York Heart Association class III or IV heart disease
* No unstable angina pectoris
* No cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No cerebrovascular accident or transient ischemic attack within the past 6 months
* No history of orthostatic hypotension
* No evidence of acute ischemia or significant conduction abnormality (left anterior hemiblock in the presence of right bundle branch block or second or third degree atrioventricular blocks) on electrocardiogram
* No uncontrolled hypertension requiring antihypertensive medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Febrile episodes up to 38.5°C allowed if no evidence of active infection
* No other uncontrolled concurrent illness
* No known or active HIV infection
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study entry
* At least 3 months since prior monoclonal antibody therapy (e.g., rituximab)
* No more than 3 prior regimens of conventional cytotoxic chemotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* At least 1 week since prior steroid therapy
* At least 4 weeks since prior radiotherapy and recovered
* At least 4 weeks since prior major surgery
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2001-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gerecitano, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 06/21/2001 Protocol Closed to Accrual 03/11/2008 Primary Completion Date 03/10/2009 Recruitment Location is the medical clinic
Groups:
- PS-341 (Bortezomib): Patients receive an infusion of bortezomib over 3-5 seconds two times a week for two weeks or once weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve at least a partial response lasting at least 6 months may receive retreatment.
Period: Overall Study
Arm/Group | PS-341 (Bortezomib)
Started | 103
Completed | 89
Not Completed | 14
Not completed — Other | 1
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Progression of disease | 6
Not completed — patient received other treatment | 1
Not completed — delay in obtaining staging images | 1

BASELINE CHARACTERISTICS:
Arm/Group | PS-341 (Bortezomib)
Number analyzed (Participants) | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 65
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The response probability will be estimated. The 95% confidence interval will be provided.
Time Frame: Up to 3 years
Measure: Number; unit: participants
Groups:
- PS-341 (Bortezomib)-Relapsed Patients; PS-341 (Bortezomib)-Refractory Patients: Patients receive an infusion of bortezomib over 3-5 seconds two times a week for two weeks or once weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve at least a partial response lasting at least 6 months may receive retreatment.
Arm/Group | PS-341 (Bortezomib)-Relapsed Patients | PS-341 (Bortezomib)-Refractory Patients
Number analyzed (Participants) | 23 | 14
participants | 11 | 6

ADVERSE EVENTS:
Arm/Group | PS-341 (Bortezomib)
Serious Adverse Events (participants affected / at risk) | 20/103
Other Adverse Events (participants affected / at risk) | 95/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS-341 (Bortezomib) (N=103)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infection, NOS (Infections and infestations) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neurological disorder (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Platelet count decrease (Investigations) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PS-341 (Bortezomib) (N=103)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Alkaline Phosphatase (Investigations) | 25 (25)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Bilirubin (Investigations) | 25 (25)
Constipation (Gastrointestinal disorders) | 22 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine (Investigations) | 24 (24)
Diarrhea (Gastrointestinal disorders) | 30 (30)
Dizziness (Nervous system disorders) | 10 (10)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Edema (General disorders) | 5 (5)
Fatigue (General disorders) | 33 (33)
Fever (General disorders) | 6 (6)
Headache (Nervous system disorders) | 7 (7)
Anemia (Hemoglobin decrease) (Blood and lymphatic system disorders) | 72 (72)
Hyperglycemia (Metabolism and nutrition disorders) | 73 (73)
Hyperkalemia (Metabolism and nutrition disorders) | 17 (17)
Hypernatremia (Metabolism and nutrition disorders) | 19 (19)
Hypoalbuminemia (Metabolism and nutrition disorders) | 38 (38)
Hypocalcemia (Metabolism and nutrition disorders) | 37 (37)
Hypoglycemia (Metabolism and nutrition disorders) | 11 (11)
Hypokalemia (Metabolism and nutrition disorders) | 13 (13)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 27 (27)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (11)
Insomnia (Psychiatric disorders) | 5 (5)
White blood cell decrease (Investigations) | 51 (51)
Lymphocyte count decreased (Investigations) | 41 (41)
Nausea (Gastrointestinal disorders) | 25 (25)
Neuropathy-peripheral (Nervous system disorders) | 14 (14)
Neuropathy-sensory (Nervous system disorders) | 39 (39)
Neutrophil count decreased (Investigations) | 43 (43)
PT (Investigations) | 11 (11)
PTT (Investigations) | 10 (10)
Pain, other (General disorders) | 7 (7)
Platelet count decrease (Investigations) | 84 (84)
Rash (Skin and subcutaneous tissue disorders) | 11 (11)
Rigors, chills (General disorders) | 6 (6)
Aspartate aminotransferase increase (Investigations) | 34 (34)
Alanine aminotransferase increase (Investigations) | 28 (28)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 12 (12)
Weight loss (Investigations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less